CLINICAL TRIAL: NCT07258966
Title: The Effect of Integrating Transtheoretical Model in Contraceptive Methods Training on University Students: A Randomized Control Trial
Brief Title: Contraception Training Using the Transtheoretical Model in Students (CT-TTM)
Acronym: CT-TTM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Near East University, Turkey (Other)
Responsible Party: Principal Investigator, Jonathan Nicıza, Principal Investigator, Near East University, Turkey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: neu/2025/001
Record Dates: First submitted 2025-10-02; First posted 2025-12-02 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Contraception; Health Behavior
Keywords: Transtheoretical Model; Contraception; Contraceptive Methods Training; University Students; Health Behavior Change; Reproductive Health; Randomized Controlled Trial; Unsafe Sexual Behavior
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Intervention Model Description: Participants are assigned to either the TTM training or the control group and remain there. This confirms the use of random assignment to create the intervention and control groups, but the intervention is for the treatment group. the control group receive no specific program.
Masking Description: The only party that could potentially have been masked was the Outcomes Assessor; however, the study protocol dictated no party was formally blinded to simplify data collection and management
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transtheoretical Model (TTM) Contraceptive Training (Experimental): The material was included a PowerPoint presentation, educational videos, and scientific articles to enhance learning. Each session lasted 60 minutes and was held once a week over seven weeks; one topic was covered in each session. The integration of the TTM framework was systematically applied throughout the contraception education program.
  Interventions: Other: Contraceptive method training

INTERVENTIONS:
Other: Contraceptive method training — The intervention is to determine the effect of the TTM intervention on nursing student knowledge, attitude and behavior towards contraceptive method. The study is conducted as a randomized controlled trial

SUMMARY:
What was the study about? This study tested whether a special training program based on the Transtheoretical Model (TTM) could help university students improve their knowledge, attitudes, and actual behavior related to contraception. The goal was to see if this method could reduce risky sexual behavior that leads to issues like sexually transmitted infections and unplanned pregnancies.

How was the study done? It was a high-quality study called a Randomized Clinical Trial (RCT).

* Participants: 68 international nursing students were split into two groups randomly.
* Intervention Group (34 students): Received the specialized TTM-based contraceptive training.
* Control Group (34 students): Did not receive the special training (they likely received standard care or nothing).
* Comparison: Researchers then compared the two groups to see if the training made a difference.

What will the study measure? The primary outcome is the change in the composite score of contraceptive competencies (knowledge, attitude, and behavior) one week after the intervention, comparing the Intervention Group to the Control Group.

What is the significance? This trial will determine the efficacy of a Transtheoretical Model-based intervention as a targeted strategy to improve contraceptive competencies and inform evidence-based health education for young adults.

DETAILED DESCRIPTION:
Detailed Description

1. Rationale and Background Unprotected sexual intercourse among young adults, particularly in the 15-49 age group, presents substantial public health challenges globally, resulting in high rates of sexually transmitted infections (STIs), unintended pregnancies, and induced abortions. Providing efficacious contraceptive knowledge and fostering informed decision-making are critical public health objectives, yet utilization is often hindered by sociocultural barriers such as religious convictions, community prejudices, and partner opposition.

   This study directly addresses this need by utilizing the Transtheoretical Model (TTM) of Behavior Change to design and evaluate a structured contraceptive education program targeting international nursing students. The TTM is a widely accepted, stage-based framework positing that individuals move through distinct stages (Precontemplation, Contemplation, Preparation, Action, Maintenance, Termination) when modifying a health behavior. The core scientific premise of this trial is that an educational intervention tailored to an individual's specific stage of change will be significantly more effective in promoting positive contraceptive knowledge, attitudes, and behavior than a standard, untailored approach.

   The primary objective of this randomized controlled trial is to determine the effect of a TTM-based contraceptive training program on students' knowledge, attitude, and behavior regarding contraceptive methods.
2. Study Design and Setting This is a single-center, two-arm, parallel-group, superiority, single-blind Randomized Controlled Trial (RCT). The study was conducted at the Near East University, targeting the population of international nursing students. The protocol adheres to the CONSORT 2010 guidelines for randomized trials.

   Participants who scored low (0-14) on the Contraceptive Behaviour Scale (CBS) were considered eligible to ensure the intervention targeted a population with existing behavioral deficits.
3. Participants and Allocation The target population consists of international nursing students enrolled at the Near East University.

   A total of N=68 eligible participants were enrolled. The sample size calculation, performed using G*Power 3.1.9.2 software based on a medium effect size (d=0.77) from previous TTM education trials, required n=64 participants to achieve 85% power at α=0.05. An additional 5% was added for potential attrition, yielding a final N=68 (34 per arm).

   Randomization: Simple randomization was performed using a web-based random number generator ('randomiser.org') by an expert external to the research team. The assignments were sealed in opaque envelopes. After baseline data collection (pre-test), the envelopes were opened by the researcher to assign participants to either the Intervention Group or the Control Group.

   Blinding: This was a single-blind trial, where the participants were necessarily unmasked to their group assignment due to the nature of the active educational intervention. However, the researcher who administered the follow-up tests and the statistical analyst were blinded to the group allocations.
4. Interventions

   The intervention phase consisted of two groups:

   Intervention Group This arm received a comprehensive, structured educational program consisting of seven weekly 60-minute interactive sessions. The content was reviewed by five subject matter experts (3 Public Health Nursing, 1 Obstetrics and Gynaecology Nursing, 1 Sex Therapist) and systematically integrated with the TTM framework.

   The educational content covered the necessity of contraception, common misconceptions, high fertility awareness, STIs and abortion, contraceptive method classification, effectiveness, advantages, disadvantages, and contraindications. The final session was a unique component dedicated to teaching students how to apply the TTM framework to their future clients. Throughout the seven sessions, the TTM was utilized to tailor educational strategies:

   Pre-contemplation/Contemplation: Emphasized consciousness raising, dramatic relief, and risk awareness (Sessions 2-5).

   Preparation/Action: Provided detailed counseling on method types, overcoming obstacles, and self-efficacy (Sessions 6-8).

   Maintenance: Reinforced long-term adherence and consultation behaviors. One student was excluded due to non-attendance, leaving n=33 in the final intervention arm.

   Control Group Participants in the control arm did not receive any specific, structured intervention from the research team during the intra-phase. They followed their normal university curriculum, which includes only elementary information regarding reproductive health integrated into various standard courses. This design controls for the passage of time and standard exposure to reproductive health topics.
5. Data Collection tools

   Data were collected at two phases: Pre-Phase (Baseline), Post-Phase (One week post-intervention). The specific, validated tools used for measurement were:

   Outcome Variable: Contraceptive Knowledge (Dependent), Attitude toward Contraception (Dependent), Contraceptive Behavior (Dependent) Assessment Tool: Contraceptive Knowledge Assessment Form (CKA), Contraceptive Attitude Scale (CAS), Contraceptive Behaviour Scale (CBS) Metric/Range: MCQ (0-25 score) Knowledge, 5-point Likert (32-160 score) Attitude, 5 items (0-20 score) Behaviour.

   Administration Time: Baseline, Post-Intervention.
   * Primary Dependent Variable: A composite of contraceptive competencies (knowledge, attitude, and behavior).
   * Independent Variable: The Transtheoretical Model-based training program.
6. Statistical Analysis Data analysis was performed using SPSS (version 27). Given that the Shapiro-Wilk test indicated a non-normal distribution for the variables, non-parametric statistical methods were employed.

   * Descriptive Statistics: Frequencies, percentages, medians, and interquartile ranges were calculated.
   * Within-Group Analysis: The Wilcoxon signed-rank test was used to examine changes in knowledge, attitude, and behavior scores from baseline to post-intervention within each group.
   * Between-Group Analysis: The Mann-Whitney U test was used to compare the difference in outcome measure scores between the Intervention and Control groups.
   * Significance: All tests were two-tailed with the level of significance set at α=0.05.
   * Effect Size: Effect sizes (r) were computed to quantify the magnitude of the observed differences.

   The research hypotheses H01, H02, H03 all state a null effect of the TTM-based training on knowledge, attitudes, and behaviors, respectively.
7. Ethical Oversight The study protocol received ethical approval from the Institutional Review Board (IRB) of the Near East University (Approval ID: 1891/2024/127). All procedures were conducted in compliance with the Declaration of Helsinki on Human Rights. Informed consent was obtained from all participating nursing students prior to their involvement in the study.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers within the international nursing student group
* Sexually active
* Individuals with low scores (0-14 score) on the 'Contraceptive Behaviour Scale'.

Exclusion Criteria:

* Those who do not want to participate in the study
* Those under the age of 18
* Those who are planning a pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-01-20 (Actual); Study Completion 2025-03-10 (Actual)

PRIMARY OUTCOMES:
Contraceptive Behavior Scale (CBS) | Post-Intervention (7 Weeks)
  Change in the Contraceptive Behavior Scale (CBS) total score from Baseline (Pre-test) to Post-Intervention (1 week after the 7-session training). The CBS is a 5-item scale with a score range of 0 (minimum behavior) to 20 (maximum behavior). This measure will assess the effect of the TTM-based training on participants' contraceptive behavior.

SECONDARY OUTCOMES:
Contraceptive Attitude Scale (CAS) Score | Post-Intervention (7weeks)
  Change in the total score on the Contraceptive Attitude Scale (CAS) from Baseline to Post-Intervention. The CAS is a 32-item, 5-point Likert scale with a score range of 32 (minimum attitude) to 160 (maximum attitude). Higher scores indicate a more positive attitude toward contraceptive use.
Contraceptive Knowledge Assessment (CKA) Score Change in Contraceptive Knowledge Score 2. For Attitude: Change in Attitude Score toward Contraceptive Use | Post-Intervention (7weeks)
  Change in the total score on the Contraceptive Knowledge Assessment Form (CKA) from Baseline to Post-Intervention. The CKA consists of 25 Multiple Choice Questions (MCQ) with a score range of 0 (minimum knowledge) to 25 (maximum knowledge). Higher scores indicate better contraceptive knowledge.

CONTACTS AND LOCATIONS:
Overall Officials: Umran, Prof, Principal Investigator — Near East University
Locations (1):
- Near East University Turkey, Nicosia, Cyprus

IPD SHARING:
Plan to Share IPD: No